CLINICAL TRIAL: NCT00806611
Title: A Randomized, Controlled Trial of Intraoperative Celiac Plexus Neurolysis for Patients With Operable (Resectable and Unresectable) Pancreatic and Periampullary Cancer
Brief Title: Intraoperative Celiac Plexus Neurolysis for Patients With Operable Pancreatic and Periampullary Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08D.380; 2007-32 (Other: CCRRC); JT 1239 (Other: JeffTrial Number)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; periampullary cancer; resectable; unresectable; celiac plexus neurolysis; surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50% Ethanol (Experimental): Operating surgeon injects 20 ml of 50% ethanol on each side of the aorta at the level of the celiac axis with a 20 or 22 gauge spinal needle
  Interventions: Procedure: Alcohol Block
- Placebo (Placebo Comparator): Operating surgeon injects 20 ml of saline on each side of the aorta at the level of the celiac axis with a 20 or 22 gauge spinal needle
  Interventions: Procedure: Alcohol Block

INTERVENTIONS:
Procedure: Alcohol Block — Operating surgeon by injecting 20 ml of either 50% ethanol or saline on each side of the aorta at the level of the celiac axis with a 20 or 22 gauge spinal needle
  Other Names: ethanol celiac plexus neurolysis

SUMMARY:
Determine if the addition of an intraoperative ethanol celiac plexus neurolysis (alcohol block) in patients undergoing surgical intervention for pancreatic cancer will result in a decrease in cancer associated pain

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma is the fourth leading cause of cancer related death in the United States and is usually fatal. Surgery provides the only chance for long-term survival. Pain is a significant, often difficult to control component of survivorship for many who succumb to this disease. The purpose of this trial is to evaluate the effect of ethanol celiac plexus neurolysis (alcohol nerve block) in patients undergoing surgical intervention for pancreatic cancer. Patients undergoing surgery for pancreatic cancer will be enrolled in a prospective randomized double blind placebo controlled clinical trial.

This protocol is designed to definitively determine the role of ethanol celiac plexus neurolysis as a simple addition to the surgical management of pancreatic adenocarcinoma and help define the standard of care for cancer associated pain management in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative imaging indicates possibility of resectable pancreatic cancer
* Intraoperative biopsy histologically confirming pancreatic adenocarcinoma

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is cancer related pain control. | Increased pain at 12 months in subjects with resectable tumors; increased pain at 3 months in subjects with unresectable tumors

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lavu H, Lengel HB, Sell NM, Baiocco JA, Kennedy EP, Yeo TP, Burrell SA, Winter JM, Hegarty S, Leiby BE, Yeo CJ. A prospective, randomized, double-blind, placebo controlled trial on the efficacy of ethanol celiac plexus neurolysis in patients with operable pancreatic and periampullary adenocarcinoma. J Am Coll Surg. 2015 Apr;220(4):497-508. doi: 10.1016/j.jamcollsurg.2014.12.013. Epub 2014 Dec 17. PMID 25667135
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/